CLINICAL TRIAL: NCT03317106
Title: the Prospective Study on the Incidence and the Association Between Motor Subtypes and Outcome of Delirium in Ischemic Stroke Patients
Brief Title: the Incidence and the Association Between Motor Subtypes and Outcome of Delirium in Ischemic Stroke Patients
Status: Completed | Type: Observational
Sponsor: Chungnam National University Hospital (Other)
Responsible Party: Principal Investigator, Heewon Yang, Principal Investigator, Chungnam National University Hospital
Other Study IDs: 2017-07-058
Record Dates: First submitted 2017-10-18; First posted 2017-10-23 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Delirium; Cerebral Infarction
MeSH Terms: conditions — Delirium; Cerebral Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks

SUMMARY:
this study examines the incidence of newly developed delirium in patients who admit to university hospital stroke unit for cerebral infarction, and analyze the association between delirium motor subtypes and short-term outcome in post-stroke delirium patients.

ELIGIBILITY:
Inclusion Criteria:

* All cerebral infarction patients who admit to stroke unit Chungnam National University Hospital.

Exclusion Criteria:

* Any patients who refuse to enroll the study.
* Any patients who admit to Intensive Care Unit(ICU), because ICU is well-known for precipitating delirium.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All cerebral infarction patients who admit to stroke unit Chungnam National University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 943 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
mean K-DRS-R98 score | 3 weeks
  mean score of delirium severity rating scale during follow up period. Detailed information about scale: Korean Version of the Delirium Rating Scale-Revised-98(K-DRS-R98) DRS-R98 proved to be a valid and reliable instrument for the assessment of delirium severity and distinguish patients with delirium from non-delirious patients including dementia. The scale is composed of two sections. The first section is the severity scale, which consists of 13 items that are scored from 0 to 3 according to a Likert scale that is anchored by descriptions of phe-nomenology. The second section consists of three diagnostic items that are scored from 0 to 2 or 3. These items include temporal onset of symptoms, fluctuation of symptom severity and physical disorder. The total scale is comprised of 16 items. The total score is the sum of the scores for each item and the higher the score, the greater the severity.

CONTACTS AND LOCATIONS:
Overall Officials: Jeonglan Kim, Study Chair — Professor
Locations (1):
- Chungnam National University Hospital, Daejeon, Munhwa-ro 282, Jung-gu, South Korea